CLINICAL TRIAL: NCT02744911
Title: Development of a Telehealth Platform for Treatment With the SpeechVive Device
Brief Title: Development of Software to Provide the SpeechVive Device Via the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SpeechVive, Inc (Industry)
Collaborators: Purdue University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R44DC014867-01A1 (NIH)
Record Dates: First submitted 2016-04-06; First posted 2016-04-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: speech problems
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Telemedicine group (Experimental): People with Parkinson's disease and their caregivers obtaining treatment using the SpeechVive device via the internet using the telemedicine application. Also includes speech-language pathologists providing treatment via the telemedicine application.
  Interventions: Device: SpeechVive device; Behavioral: Telemedicine interaction
- In person group (Active Comparator): People with Parkinson's disease and their caregivers obtaining treatment using the SpeechVive device in person. Also includes speech-language pathologists providing treatment in person.
  Interventions: Device: SpeechVive device; Behavioral: In person interaction

INTERVENTIONS:
Device: SpeechVive device — The SpeechVive is a wearable device that plays multi-talker babble noise in one ear while the person wearing it is talking. The noise is voice-activated (only present when the person speaks). The noise does not interfere with the ability to hear communication partners. The noise coming from the device functions as a natural external cue for people with Parkinson's disease to talk more loudly and clearly. Treatment will involve asking the participants to wear the device daily during the treatment period.
Behavioral: Telemedicine interaction — Participants will interact with the speech-language pathologist using the telemedicine platform from their home.
  Arms: Telemedicine group
Behavioral: In person interaction — Participants will interact with the speech-language pathologist in-person at the speech pathologist's office
  Arms: In person group

SUMMARY:
Telehealth, increasingly recognized in the neurology field as a solution to access issues for people with Parkinson's disease, improves access to speech therapy, particularly those living in rural areas or with travel barriers. The SpeechVive device, developed by SpeechVive, Inc., is a treatment solution that is easy to use and effective. In an NIH funded study, the SpeechVive device improved communication in 90% of individuals with PD by improving volume, articulation, and speech rate. The investigators propose to eliminate the one drawback of the SpeechVive device, namely that it currently must be programmed by a speech-language pathologist for each patient in person. The overall goal of this project is to develop a telehealth platform for the SpeechVive device that will enable video conferencing for treatment and remote programming of the SpeechVive device for each patient. Once the platform has been developed, the investigators will conduct a study to examine effectiveness and the patient and caregiver satisfaction with telepractice using the SpeechVive device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Difficulty communicating
* Is currently being seen, or agrees to be seen, by a speech pathologist who fits the SpeechVive device and also has agreed to participate in the study
* Has a regular caregiver living with him/her

Exclusion Criteria:

* Neurological diagnoses (except Parkinson's disease)
* Bilateral hearing aids (since one free ear is required for use of the SpeechVive device)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Quality of Life | Change from baseline after 6 months of treatment
  Scale of Quality of Life of Care-givers
Depression: Caregiver Geriatric Depression Scale | Change from baseline after 6 months of treatment
  Geriatric Depression Scale
Change in Patient with PD Ratings of Communication Competence | Change from baseline after 6 months of treatment
  Communicative Participation Item Bank-Short Form
Change in Patient with PD quality of life | Change from baseline after 6 months of treatment
  Parkinson's Disease Questionnaire-39
Attractiveness of the telehealth platform. | At monthly intervals during the study period (6 months for each patient)
  Survey requesting SLP data regarding patients seen during the study period and adoption of the telepractice model by patients
Travel cost burden - in-person group | At monthly intervals during the study period (6 months for each patient)
  Survey requesting Patient/caregiver travel distances and durations
Impact of treatment on time - telemedicine group | At monthly intervals during the study period (6 months for each patient)
  Survey requesting Patient and caregiver reports of time spent before and after sessions preparing and setting up equipment and clearing equipment
Treatment adherence | At monthly intervals during the study period (6 months for each patient)
  Usage data from the SpeechVive and patient attendance at treatment sessions
Change in Vocal intensity level | Change from baseline after 6 months of treatment
  Sound pressure level from speech samples with and without the device in place
Change in Patient with PD Depression Level | Change from baseline after 6 months of treatment
  Geriatric Depression Scale Short form
Impact of Life Events for Patient with PD and Caregiver | Change from baseline after 6 months of treatment
  Change in Impact of PD on life satisfaction
Change in general self-efficacy | Change from baseline after 6 months of treatment
  Self-efficacy for people with disabilities scale

SECONDARY OUTCOMES:
Change in Speech rate | Change from baseline after 6 months of treatment
  Rate of speech from speech samples with and without the device in place
Change in Pausing patterns | Change from baseline after 6 months of treatment
  Number and duration of silent and filled pauses from speech samples with and without the device in place
Change in Caregiver Burden | Change from baseline after 6 months of treatment
  Caregiver Burden Inventory
Change in Apathy | Change in baseline after 6 months of treatment for Patient with PD and Caregiver
  Apathy Scale
Change in Caregiver Ratings Patient's of Communication Competence | Change in baseline after 6 months of treatment
  Communicative Participation Item Bank-Short Form
Change in Patient with PD Participation in Social Activities | Change in baseline after 6 months of treatment
  Quality of Life in Neurological Disorders (Neuro-QOL)
Change in Patient with PD Participation in Social Activities | Change in baseline after 6 months of treatment
  Ability to Participate in Social Roles and Activities-Short Form
Change in Patient with PD Perceived Autonomy | Change in baseline after 6 months of treatment
  7-item Autonomy Subscale of the Basic Psychological Needs Scale
Patient with PD satisfaction - telemedicine group | At the end of the study period (after 6 months)
  Survey requesting ratings of satisfaction with the telemedicine application and treatment process
Caregiver satisfaction - telemedicine group | At the end of the study period (after 6 months)
  Survey requesting ratings of satisfaction with the telemedicine application and treatment process
Patient with PD satisfaction - in person group | At the end of the study period (after 6 months)
  Survey requesting ratings of satisfaction with the in-person treatment process
Caregiver satisfaction - in person group | At the end of the study period (after 6 months)
  Survey requesting ratings of satisfaction with the in-person treatment process

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - SpeechVive, Inc, Lafayette, Indiana
  - Purdue University, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: Yes
The data from the people with Parkinson's disease and their caregivers will include limited financial information, perceptions of speech telepractice, survey data, and some objective measurements of speech production. Once de-identified and published in peer-reviewed journals, these data will be made available upon request. Any researcher requesting access to these data will need to submit the following to Jessica Huber:
  1. Name and institution of PI
  2. Proof of institutional appointment
  3. Names and roles for all individuals who will access the data for the planned analysis
  4. Detailed plan for the use of the data
  5. Timeline for use and publication of the analyses If Dr. Huber approves the data use, the PI must sign a license with Purdue University's Office of Technology Commercialization promising to keep the data confidential, to not share it with anyone not named in the application above, and to destroy the data once analysis is complete.

REFERENCES:
- [Background] Stathopoulos ET, Huber JE, Richardson K, Kamphaus J, DeCicco D, Darling M, Fulcher K, Sussman JE. Increased vocal intensity due to the Lombard effect in speakers with Parkinson's disease: simultaneous laryngeal and respiratory strategies. J Commun Disord. 2014 Mar-Apr;48:1-17. doi: 10.1016/j.jcomdis.2013.12.001. Epub 2013 Dec 28. PMID 24438910
- [Background] Huber JE, Darling M, Francis EJ, Zhang D. Impact of typical aging and Parkinson's disease on the relationship among breath pausing, syntax, and punctuation. Am J Speech Lang Pathol. 2012 Nov;21(4):368-79. doi: 10.1044/1058-0360(2012/11-0059). Epub 2012 Jul 30. PMID 22846880
- [Background] Darling M, Huber JE. Changes to articulatory kinematics in response to loudness cues in individuals with Parkinson's disease. J Speech Lang Hear Res. 2011 Oct;54(5):1247-59. doi: 10.1044/1092-4388(2011/10-0024). Epub 2011 Mar 8. PMID 21386044
- [Background] Huber JE, Darling M. Effect of Parkinson's disease on the production of structured and unstructured speaking tasks: respiratory physiologic and linguistic considerations. J Speech Lang Hear Res. 2011 Feb;54(1):33-46. doi: 10.1044/1092-4388(2010/09-0184). Epub 2010 Sep 15. PMID 20844256
- [Background] Sadagopan N, Huber JE. Effects of loudness cues on respiration in individuals with Parkinson's disease. Mov Disord. 2007 Apr 15;22(5):651-9. doi: 10.1002/mds.21375. PMID 17266087